CLINICAL TRIAL: NCT04178733
Title: A Single-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of LY3493269 in Healthy Participants
Brief Title: A Safety Study of LY3493269 Given as a Single Injection in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17452; J1X-MC-GZHA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo - SC (Placebo Comparator): Participants received Placebo subcutaneously (SC).
  Interventions: Drug: Placebo - SC
- 0.5 mg LY3493269 IV (Experimental): Participants received 0.5 mg LY3493269 intravenously (IV).
  Interventions: Drug: LY3493269 - IV
- 0.15 mg LY3493269 SC (Experimental): Participants received 0.15 mg LY3493269 SC.
  Interventions: Drug: LY3493269 - SC
- 0.5 mg LY3493269 SC (Experimental): Participants received 0.5 mg LY3493269 SC.
  Interventions: Drug: LY3493269 - SC
- 1.5 mg LY3493269 SC (Experimental): Participants received 1.5 mg LY3493269 SC.
  Interventions: Drug: LY3493269 - SC

INTERVENTIONS:
Drug: LY3493269 - SC — Administered SC
  Arms: 0.15 mg LY3493269 SC; 0.5 mg LY3493269 SC; 1.5 mg LY3493269 SC
Drug: Placebo - SC — Administered SC
  Arms: Placebo - SC
Drug: LY3493269 - IV — Administered IV
  Arms: 0.5 mg LY3493269 IV

SUMMARY:
This study is being conducted to determine the side effects related to LY3493269 given as a single injection to healthy participants. Blood tests will be performed to check how much LY3493269 gets into the bloodstream and how long the body takes to get rid of it. Each enrolled participant will receive a single dose of LY3493269 or placebo. The study will last up to approximately 71 days for each participant, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female who cannot get pregnant
* Have a body mass index (BMI) between 19 and 40 kilograms per square meter (kg/m²), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG, heart tracing), blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for ease of blood sampling

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously completed or withdrawn from this study
* Smoke more than the equivalent of 10 cigarettes per day and are unwilling to stop smoking during the inpatient stay in the study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Have been treated with weight loss medications within 3 months of screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo SC: Participants received Placebo subcutaneously (SC).
- 0.15 mg LY3493269 SC: Participants received 0.15 milligrams (mg) LY3493269 SC.
Period: Overall Study
Arm/Group | Placebo SC | 0.15 mg LY3493269 SC | 0.5 mg LY3493269 SC | 0.5 mg LY3493269 IV | 1.5 mg LY3493269 SC
Started | 6 | 6 | 6 | 7 | 8
Received at Least One Dose of Study Drug | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 1 | 2
Not completed — Investigator Decision | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo SC: Participants received Placebo subcutaneously(SC).
- Total: Total of all reporting groups
Arm/Group | Placebo SC | 0.15 mg LY3493269 SC | 0.5 mg LY3493269 SC | 0.5 mg LY3493269 IV | 1.5 mg LY3493269 SC | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.9) | 40.8 (8.6) | 43.5 (8.5) | 36.5 (12.7) | 34.7 (9.9) | 40.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 6 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 6 | 6 | 6 | 6 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Time Frame: Baseline through final follow-up (Up To Day 43)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | 0.15 mg LY3493269 SC | 0.5 mg LY3493269 SC | 0.5 mg LY3493269 IV | 1.5 mg LY3493269 SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time Zero to Infinity (AUC 0-∞) of LY3493269
Description: Pharmacokinetics (PK): Area Under the Concentration time curve from time zero to infinity (AUC 0-∞) of LY3493269
Time Frame: Day 1: Predose, 6, 12 hours; Day 2: 24 hours; Day 3: 48 hours; Day 4: 72 hours; Day 5: 96 hours; Day 6:120 hours; Day 8:168 hours; and any time during the visit on Day 15, Day 29, Day 43 and early termination
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 0.15 mg LY3493269 SC | 0.5 mg LY3493269 SC | 0.5 mg LY3493269 IV | 1.5 mg LY3493269 SC
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanograms*hour per milliliter (ng*h/mL) | 4990 (26) | 21800 (24) | 24600 (23) | 7300 (21)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3493269
Description: PK: Maximum Concentration (Cmax) of LY3493269
Time Frame: Day 1: Predose, 6, 12 hours; Day 2: 24 hours; Day 3: 48 hours; Day 4: 72 hours; Day 5: 96 hours; Day 6:120 hours; Day 8:168 hours; and any time during the visit on Day 15, Day 29, Day 43 early termination
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.15 mg LY3493269 SC | 0.5 mg LY3493269 SC | 0.5 mg LY3493269 IV | 1.5 mg LY3493269 SC
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 16.4 (19) | 68.8 (40) | 181 (15) | 247 (27)

4. Secondary Outcome: PK: Time to Maximum Concentration (Tmax) of LY3493269
Description: PK: Time to Maximum Concentration (Tmax) of LY3493269
Time Frame: as for outcome 3
Population: All participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | 0.15 mg LY3493269 SC | 0.5 mg LY3493269 SC | 0.5 mg LY3493269 IV | 1.5 mg LY3493269 SC
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours (hr) | 12.01 [6.00 to 96.73] | 12.06 [12.00 to 96.00] | 0.39 [0.25 to 2.00] | 12.00 [12.00 to 96.08]

ADVERSE EVENTS:
Time Frame: Baseline Up To 43 Days
Description: All participants who received at least one dose of study drug.
Groups:
- Placebo SC: Participants received Placebo SC.
- 0.5 mg LY3493269 IV: Participants received 0.5 mg LY3493269 IV.
Arm/Group | Placebo SC | 0.15 mg LY3493269 SC | 0.5 mg LY3493269 SC | 0.5 mg LY3493269 IV | 1.5 mg LY3493269 SC
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 6/6 | 6/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SC (N=6) | 0.15 mg LY3493269 SC (N=6) | 0.5 mg LY3493269 SC (N=6) | 0.5 mg LY3493269 IV (N=6) | 1.5 mg LY3493269 SC (N=6)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (4) | 5 (6) | 3 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (8)
Catheter site bruise (General disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site erosion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 5 (5) | 5 (6)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 3 (5)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT04178733/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04178733/SAP_001.pdf